CLINICAL TRIAL: NCT04092972
Title: Safety and Efficacy of Interventional Treatment Through Atherectomy to Improve Vascular Functions and Patency in Symptomatic Peripheral Artery Disease - Pilot Study
Brief Title: Safety and Efficacy of Atherectomy on VasculaR Functions
Acronym: SAVioR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Collaborators: Straub Medical AG (Industry)
Responsible Party: Principal Investigator, Fadi Al-Rashid, MD, Principal Investigator, University Hospital, Essen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SAVioR_CR
Record Dates: First submitted 2019-04-17; First posted 2019-09-17 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease; Claudication, Intermittent
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Atherectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atherectomy (Experimental): Atherectomy and drug-coated balloon (DCB)
  Interventions: Other: Atherectomy
- Standard care (Active Comparator): Standard care with predilation (POBA) and DCB
  Interventions: Other: POBA and DCB

INTERVENTIONS:
Other: Atherectomy — Straub Rotarex S atherectomy and drug-coated balloon DCB. Predilation of the lesion with a predefined ballon (180 sec, Passeo-18). Thus, no direct DCB will be conducted. All DCB lengths (40mm to 200 mm) and Diameters (3mm to 7mm) are eligible for the Trial as long as used in the superficial femoral artery (SFA).
  Arms: Atherectomy
Other: POBA and DCB — Standard predilation (POBA) and DCB. Predilation of the lesion with a predefined ballon (180 sec, Passeo-18). Thus, no direct DCB will be conducted. All DCB lengths (40mm to 200 mm) and Diameters (3mm to 7mm) are eligible for the Trial as long as used in the superficial femoral artery (SFA).
  Arms: Standard care

SUMMARY:
Interventional strategies aim to restore tissue perfusion. However, despite the simple reopening of a narrowed artery they affect endothelial function, perpetuating dysfunctional vascular homeostasis. PTA and atherectomy might alter the endothelial function but the mechanisms are incompletely understood. The primary goal of atherectomy is vessel preparation and improving compliance, which could aid in preserving vessel functions. Aim of this study is to determine safety, efficacy, patency and vessel functions in the femoropopliteal artery following atherectomy and DCB.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease, lesions in the SFA and popliteal artery.
* Clinical diagnosis of chronic, symptomatic lower limb ischemia as defined by Rutherford 2, 3, or 4
* Planed peripheral intervention TASC A-D
* Subject must be between 18 and 85 years old
* Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12-month angiographic evaluation
* Vessel diameter ≥3.0 mm and ≤7.0 mm
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures

Exclusion Criteria:

* Thrombolysis within 72 hours prior to the index procedure
* Aneurysm in the femoral artery or popliteal artery
* Concomitant hepatic insufficiency, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Unstable angina pectoris at the time of the enrollment
* Recent myocardial infarction or stroke < 30 days prior to the index procedure
* Life expectancy less than 12 months
* Septicemia at the time of enrollment
* Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb
* Known or suspected allergies or contraindications to aspirin, clopidogrel or heparin Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-28 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-Emerged Adverse Events | 6 months Follow Up
  Incidence of Treatment-Emerged Adverse Events as assessed by angiography and adverse event assessment
Primary patency | 6 months Follow Up
  determined through doppler ultrasound

SECONDARY OUTCOMES:
Bail-out stent rate | 6 months Follow Up
  success of atherectomy in the SFA including the bail-out stenting rates
FMD local | 6 months Follow Up
  Local endothelial function and vasomotion testing as determinded by FMD of the femoral artery
Vessel stiffness | 6 months Follow Up
  Vascular stiffness determined through pulse wave velocity (PWV)
target lesion revascularization | 6 months Follow Up
  freedom from Target Lesion Revascularization (FTLR) is defined as the Need for percutaneous or interventional revascularization
ABI (Ankle Brachial Index) | 6 months Follow Up
  Ankle Brachial Index assessed by Doppler
Systemic endothelial function | 6 months Follow Up
  Change of endothelial function, assessed by the change in the vasodilation after reactive hyperaemia of the brachial artery (flow-mediated dilation = FMD)
Change in Plaque burden | during baseline visit
  Change in plaque burden is measured by plaque volume change using intravascular ultrasound (IVUS)
Change in plaque characteristic | during baseline visit
  Change in plaque characteristic is quantified using virtual histology using intravascular ultrasound (IVUS)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Rammos, Principal Investigator — Universität Duisburg-Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rammos C, Manzke A, Lortz J, Messiha D, Petrikhovich O, Janosi RA, Steinmetz M, Rassaf T. Mechanical atherothrombectomy improves endothelial function through plaque burden reduction in PAD. Vasa. 2022 Nov;51(6):377-385. doi: 10.1024/0301-1526/a001034. Epub 2022 Oct 4. PMID 36193630